CLINICAL TRIAL: NCT03103438
Title: An Open-Label, Dose Escalation Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of a Single Subcutaneous Dose of BCD-089 in Healthy Volunteers
Brief Title: First-in-human Study of Safety, Pharmacokinetics and Pharmacodynamics of Various Doses of BCD-089 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: BCD-089-1
Record Dates: First submitted 2017-03-24; First posted 2017-04-06 (Actual); Results first posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Healthy
MeSH Terms: interventions — levilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Cohort 1 (Experimental): his cohort includes one subject who will receive the maximum safe starting dose of BCD-089 (0.06 mg/kg) subcutaneously. If the dose limitating toxicity occurs within the first seven days after injection the study will be stopped. If there is no DLT within mentioned above period then Cohort no.2 is included.
  Interventions: Biological: BCD-089
- Cohort 2 (Experimental): This cohort includes 3 subjects who will receive the single subcutaneous injection of BCD-089 at a dose of 0.3 mg/kg.If at least 2 subjects are observed to have DLT, this dose level is defined as the MTD (unless only 3 patients have been treated at that level, in which case it is the tentative MTD). If 0 of the 3 subjects are observed to have DLT, the dose level is escalated one step for the next cohort no.3 of 3 subjects, and the process continues as above. If exactly 1 of the 3 subjects treated show DLT, 3 additional subjects are treated at the current dose level. If none of these additional 3 patients show DLT, the dose level is escalated for the next Cohort no. 3.
  Interventions: Biological: BCD-089
- Cohort 3 (Experimental): This cohort includes 3 subjects who will receive the single subcutaneous injection of BCD-089 at a dose of 0.625 mg/kg.If at least 2 subjects are observed to have DLT, this dose level is defined as the MTD (unless only 3 patients have been treated at that level, in which case it is the tentative MTD). If 0 of the 3 subjects are observed to have DLT, the dose level is escalated one step for the next cohort no. 4 of 3 subjects, and the process continues as above. If exactly 1 of the 3 subjects treated show DLT, 3 additional subjects are treated at the current dose level. If none of these additional 3 patients show DLT, the dose level is escalated for the next Cohort no. 4.
  Interventions: Biological: BCD-089
- Cohort 4 (Experimental): This cohort includes 3 subjects who will receive the single subcutaneous injection of BCD-089 at a dose of 1.0 mg/kg. If at least 2 subjects are observed to have DLT, this dose level is defined as the MTD (unless only 3 patients have been treated at that level, in which case it is the tentative MTD). If 0 of the 3 subjects are observed to have DLT, the dose level is escalated one step for the next cohort no. 5 of 3 subjects, and the process continues as above. If exactly 1 of the 3 subjects treated show DLT, 3 additional subjects are treated at the current dose level. If none of these additional 3 patients show DLT, the dose level is escalated for the next Cohort no. 5.
  Interventions: Biological: BCD-089
- Cohort 5 (Experimental): This cohort includes 3 subjects who will receive the single subcutaneous injection of BCD-089 at a dose of 1.6 mg/kg. If at least 2 subjects are observed to have DLT, this dose level is defined as the MTD (unless only 3 patients have been treated at that level, in which case it is the tentative MTD). If 0 of the 3 subjects are observed to have DLT, the dose level is escalated one step for the next cohort no. 6 of 3 subjects, and the process continues as above. If exactly 1 of the 3 subjects treated show DLT, 3 additional subjects are treated at the current dose level. If none of these additional 3 patients show DLT, the dose level is escalated for the next Cohort no. 6.
  Interventions: Biological: BCD-089
- Cohort 6 (Experimental): This cohort includes 3 subjects who will receive the single subcutaneous injection of BCD-089 at a dose of 2.2 mg/kg. If at least 2 subjects are observed to have DLT, this dose level is defined as the MTD (unless only 3 patients have been treated at that level, in which case it is the tentative MTD). If 0 of the 3 subjects are observed to have DLT, the dose level is escalated one step for the next cohort no. 7 of 3 subjects, and the process continues as above. If exactly 1 of the 3 subjects treated show DLT, 3 additional subjects are treated at the current dose level. If none of these additional 3 patients show DLT, the dose level is escalated for the next Cohort no. 7.
  Interventions: Biological: BCD-089
- Cohort 7 (Experimental): This cohort includes 3 subjects who will receive the single subcutaneous injection of BCD-089 at a dose of 2.9 mg/kg. If at least 2 subjects are observed to have DLT, this dose level is defined as the MTD (unless only 3 patients have been treated at that level, in which case it is the tentative MTD). If exactly 1 of the 3 subjects treated show DLT, 3 additional subjects are treated at the current dose level.
  Interventions: Biological: BCD-089

INTERVENTIONS:
Biological: BCD-089
  Other Names: human monoclonal antibody to interleukin-6 receptor

SUMMARY:
This is an open label, phase 1, "3+3" dose escalating study of tolerability, safety, pharmacokinetics, pharmacodynamics and immunogenicity of a single subcutaneous injection of the novel monoclonal antibody against the interleukin-6 receptor - BCD-089. The study will enroll 19 healthy male volunteers.

DETAILED DESCRIPTION:
IL-6 is a new potential therapeutic target which plays important role in pathogenesis of several autoimmune disorders including rheumatoid arthritis. BCD-089 is a novel fully human monoclonal antibody against the interleukin-6 receptor developed by JCS BIOCAD (Russia) which is now on the first step of clinical evaluation. BCD-089-1 study is the first-in-human clinical trial which is intended to evaluate tolerability, safety, pharmacokinetics, pharmacodynamics and immunogenicity of BCD-089 when used as a single step-by-step escalating subcutaneous dose in healthy male volunteers. During this study it is expected to determine diapason of safety doses of BCD-089 (incl. MTD) which thereafter can be evaluated in phase 2 studies.

ELIGIBILITY:
Inclusion Criteria:

* singed informed consent
* male gender
* 18-45 years of age inclusively
* BMI between18.5-30.0 kg/sq.m.
* absence of any sings of hepatic, renal, gastrointestinal, cardiovascular, endocrine, respiratory, immunologic, hematologic, dermatologic, or neurologic abnormality at screening or/and in anamnesis
* parameters of complete blood count, blood biochemistry, and urinalysis do not exceed reference values, which are used at Study site laboratory
* normal hemodynamic parameters :
* absence of chronic infections (HIV, syphilis, hepatitis В or С, tuberculosis ) and chronic inflammation
* absence of infections within 4 weeks before screening
* absence of mental disorders or other conditions, which may affect the ability of participant to follow Protocol
* absence of alcohol or drug addiction signs (incl. history of such addiction).
* volunteer's ability to follow Protocol procedures
* consent of volunteers and their sexual partners with childbearing potential to use adequate contraception during screening period and the main study part (14 days before randomization and 70 day after SC injection). This requirement is not applicable in surgically sterilized volunteers. Adequate contraception includes the use of one barrier method in combination with spermicides, intrauterine device / oral contraceptives in sexual partner

Exclusion Criteria:

* history of use of monoclonal antibodies against IL-6 or IL-6R
* known severe allergy (anaphylaxis or multidrug intolerance)
* known intolerance to medicines containing monoclonal antibodies (murine, humanized, human) or to any excipients of BCD-089
* major surgery within 30 days prior screening
* severe infections (required hospitalization, parenteral use of antimicrobial agents) within 6 months prior the date of BCD-089 injection
* systemic use of antimicrobials within 2 months prior the date of BCD-089 injection
* more than 4 episodes of respiratory tract infections within 6 months prior the screening examination
* presence of any disorders which may affect pharmacokinetics of BCD-089
* history of fever which was equal or exceeded 40 degrees in Celsius
* - actual or prior depression, suicidal tendencies
* use of any medicines, vitamins, biologically active additives within 14 days prior the screening examination use of any medicines which affects hemodynamics or hepatic function within 30 days prior the screening examination simultaneous participation in any other clinical trial, as well as former participation in other clinical trials within 2 months before this study initiation.

previous participation in this study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- LLC BioEk, Saint Petersburg, Russia

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: One subject received the maximum safe starting dose of BCD-089 (0.06 mg/kg) subcutaneously.
- Cohort 2: Three subjects received the single subcutaneous injection of BCD-089 at a dose of 0.3 mg/kg.
- Cohort 3: Three subjects received the single subcutaneous injection of BCD-089 at a dose of 0.625 mg/kg.
- Cohort 4: Three subjects received the single subcutaneous injection of BCD-089 at a dose of 1.0 mg/kg.
- Cohort 5: Three subjects received the single subcutaneous injection of BCD-089 at a dose of 1.6 mg/kg.
- Cohort 6: Three subjects received the single subcutaneous injection of BCD-089 at a dose of 2.2 mg/kg.
- Cohort 7: Three subjects received the single subcutaneous injection of BCD-089 at a dose of 2.9 mg/kg.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7
Started | 1 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 1 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Total
Number analyzed (Participants) | 1 | 3 | 3 | 3 | 3 | 3 | 3 | 19
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 25 [25 to 25] | 28 [24 to 28] | 22 [22 to 22] | 23 [22 to 23] | 27 [26 to 27] | 22 [22 to 22] | 26 [24 to 26] | 25 [22 to 27]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 1 | 3 | 3 | 3 | 3 | 3 | 3 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 1 | 3 | 3 | 3 | 3 | 3 | 3 | 19
Region of Enrollment [Number; unit: participants]
  Russia | 1 | 3 | 3 | 3 | 3 | 3 | 3 | 19

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration of BCD-089-time Curve From Zero (0) Hours to 1680 Hours After the Single Subcutaneous Injection of BCD-089
Description: Area Under the Plasma Concentration of BCD-089-time Curve From Zero (0) Hours to 1680 Hours After the Single Subcutaneous Injection of BCD-089.
Time Frame: 70 days
Population: The pharmacokinetic analysis population included the data from all volunteers included in the study (n = 19).
Measure: Median (Inter-Quartile Range); unit: ng/ml*h
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7
Number analyzed (Participants) | 1 | 3 | 3 | 3 | 3 | 3 | 3
ng/ml*h | 0 [0 to 0] | 15567.9 [8364.0 to 18664.2] | 44568.6 [14441.2 to 50635.4] | 588202.2 [160711.0 to 1044464.2] | 1208489.2 [777536.3 to 1352794.3] | 4190342.2 [3891917.6 to 6676172.8] | 10512592.4 [8628174.9 to 10759494.4]

ADVERSE EVENTS:
Time Frame: 71 days from the moment of injection
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/1 | 1/3 | 1/3 | 1/3 | 0/3 | 2/3 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=1) | Cohort 2 (N=3) | Cohort 3 (N=3) | Cohort 4 (N=3) | Cohort 5 (N=3) | Cohort 6 (N=3) | Cohort 7 (N=3)
AST decreased (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
total bilirubin increased (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 1 (1)
creatinine decreased (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT03103438/Prot_SAP_000.pdf